CLINICAL TRIAL: NCT04220333
Title: Randomized Control Trial on Mandalas of Emotions
Acronym: ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Gabriela Salim Spagnol, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 64276116400005404
Record Dates: First submitted 2019-12-19; First posted 2020-01-07 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: The team, composed of five researchers, was divided in two groups: three researchers performed the interview before and after the intervention, two others applied the intervention, which divided participants in two groups: "control" and "intervention", assuming the confidentiality of this classification, as expected in a randomized, case control, blind assessment of outcome study.
  Both groups received the same initial recommendations: 'please, lie down, relax and pay attention to your breath'. The total procedure time was the same for both groups.
Who Masked: Investigator
Masking Description: The team, composed of five researchers, was divided in two groups: three researchers performed the interview before and after the intervention, two others applied the intervention, which divided participants in two groups: "control" and "intervention", assuming the confidentiality of this classification, as expected in a randomized, case control, blind assessment of outcome study.
  Both groups received the same initial recommendations: 'please, lie down, relax and pay attention to your breath'. The total procedure time was the same for both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participants received the instruction: 'please, lie down, relax and pay attention to your breath'. This procedure was carried during 15 minutes. Soon after the experiment, individual assessment was performed blinded to who received intervention using a structured questionnaire and Likert-scales about the degree of relaxation and feelings.
  Interventions: Behavioral: Control
- Intervention (Experimental): The intervention protocol was divided in two steps: first, patients spent 5 minutes in the phase of harmonization with five colored stones of a size of a walnut (green, red, yellow, white and black) placed around their bodies.
  Second, in accordance to the emotion chosen by the participant, a matching mandala was placed next to the feet, on the abdomen, or next to the head depending on the self-perceived personality type, intuitive, emotive and rational for the remaining 10 minutes (Figure 3B). The researcher also checked the control subjects once during the 15 fifteen minutes of experiment.
  Soon after the experiment, individual assessment was performed blinded to who received intervention using a structured questionnaire and Likert-scales about the degree of relaxation and feelings.
  Interventions: Behavioral: Mandalas of Emotions

INTERVENTIONS:
Behavioral: Mandalas of Emotions — Application of mandalas during 15 minutes
  Arms: Intervention
Behavioral: Control — Participants were requested to "lie down, relax and pay attention to your breath".
  Arms: Control

SUMMARY:
Epilepsy is a chronic disease with a psychosocial impact on the patient. The technique called 'Mandala of Emotions' (ME), derived from the Traditional Chinese Medicine, facilitates expression and awareness of emotions. In our pilot case study, the group "intervention with ME" managed to arouse their emotions and after the intervention felt lighter and relaxed at a higher frequency than the control group. We conducted a blind case control study to further assess usefulness of ME. Materials and Methods: Patients and caregivers recruited at an Epilepsy Outpatients Clinic with the approval of Ethics Committee were randomly divided into groups 'Control' (n=57) and 'Intervention' (n=53). In the ME group, five colored stones (green, red, yellow, white and black) were applied according to the emotion chosen by the participant. Individual assessment performed blinded to who received intervention applied a structured questionnaire and Likert-scales about the degree of relaxation and feelings pre- and post-experiment.

DETAILED DESCRIPTION:
Patients and caregivers were recruited at an Epilepsy Outpatients Clinic. This study has approval of local Ethics Committee. Participants were invited to this research at the Outpatient clinic waiting room, and when they expressed interest, they were referred to the research team. Inclusion criteria for this study were: men and women treated in the epilepsy outpatient clinic, aged 18-60 years. Volunteers signed the informed consent to participate in the study, answered a questionnaire with information about demographics, epilepsy history (age of onset, frequency, last seizure, medications). They described their emotional characteristics (intuitive, emotive, and rational) and how they felt at that moment. They were invited to choose an emotion from a list (Concern/obsession, Anger/irritation, Fear, Compassion, Sadness, Comprehension, Euphoria, Gratitude, Joy, Peace) to work on during the intervention. After, they were randomly divided into two groups: 'Control' and 'Intervention' (see Figure 1).

The Mandalas of Emotions refers to five colors in accordance to the five stages or seasons (spring, summer, high summer, fall, winter). These establish a relation to the five functional systems (liver, heart, spleen and pancreas, lungs and kidney), and to five emotions (anger, joy/euphoria, concern/obsession, sadness/melancholy, fear) with its opposite correspondents (understanding, compassion, gratitude, enthusiasm, harmony) (Ling, 2013).

Figure 1. Research procedures.

The team, composed of five researchers, was divided in two groups: three researchers performed the interview before and after the intervention, two others applied the intervention, which divided participants in two groups: "control" and "intervention", assuming the confidentiality of this classification, as expected in a randomized, case control, blind assessment of outcome study.

Both groups received the same initial recommendations: 'please, lie down, relax and pay attention to your breath'. The total procedure time was the same for both groups.

The intervention protocol was divided in two steps: first, patients spent 5 minutes in the phase of harmonization with five colored stones of a size of a walnut (green, red, yellow, white and black) placed around their bodies.

Second, in accordance to the emotion chosen by the participant, a matching mandala was placed next to the feet, on the abdomen, or next to the head depending on the self-perceived personality type, intuitive, emotive and rational for the remaining 10 minutes. The researcher also checked the control subjects once during the 15 fifteen minutes of experiment.

Soon after the experiment, individual assessment was performed blinded to who received intervention using a structured questionnaire and Likert-scales about the degree of relaxation and feelings.

Statistical analysis We first divided the groups and analyzed whether they differed in regard to sex, age, years of schooling, age of onset of seizures, time of last seizure, frequency of seizures per month, use of monotherapy and seizure control. Statistical analysis was conducted with SPSS using non-parametric tests (Mann-Whitney, ANOVA for repeated measures) and Chi-square. Content of patients perceptions were analyzed according to themes and compared between groups (control vs. intervention).

ELIGIBILITY:
Inclusion Criteria:

* men and women treated in the epilepsy outpatient clinic, aged 18-60 years. Volunteers signed the informed consent to participate in the study, answered a questionnaire with information about demographics, epilepsy history (age of onset, frequency, last seizure, medications).

Exclusion Criteria:

* Associated clinical conditions that prevented full comprehension of research procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Pre procedure Likert scale report | 15 minutes
  Before the procedure, researchers asked "How are you feeling?" and participants replied in a Likert scale from 1-Very bad to 5-Very good.
Perception of changes after 5 min of procedure | 5 minutes
  Five minutes after the procedure began, researchers applied the question: "How are you feeling?" and the researcher registered as they reported physical and emotional changes. No further measures or questionnaires were applied at this point.
Post procedure Likert scale report and qualitative questions | 15 minutes
  After the procedure, researchers asked "How are you feeling?" and participants replied in a Likert scale from 1-Very bad to 5-Very good. Researchers also applied a questionnaire with these questions: "Did you experience body changes / retrieval of memories / retrieval of specific images? Do you have any observations regarding the procedure? Researchers registered yes/no reply and participants description of changes. No further measures or questionnaires were applied after this procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroimaging Laboratory, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.